CLINICAL TRIAL: NCT01628224
Title: Enhanced Critical Care Air Transport Team Training for Mitigation of Task Saturation
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: United States Air Force (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Pritts-2010-01
Record Dates: First submitted 2011-11-18; First posted 2012-06-26 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Task Saturation
Keywords: Task saturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CCATT Team: Measurements will be taken on groups of 3 people each. There will be a total of 16 such teams, with total membership of 48 individuals

SUMMARY:
This study involves two tasks. The first involves observation of patient care during simulated aeroevacuation missions in order to gauge task saturation. The second involves review of records from actual evacuation flights in order to determine the effects of task saturation on patient care.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in a US Air Force CCATT Advanced Class at University Hospital, Cincinnati

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The population for the first task will consist of 4 CCATT teams (of 3 members each)
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Incidence of task saturation | 1 hour
  Task saturation is defined as the point at which the volume or complexity of events exceeds the capability of the individual or team to maintain a standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Pritts, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University Hospital, Cincinnati, Ohio, United States